CLINICAL TRIAL: NCT02028715
Title: Efficacy of IV Acetaminophen for Pain Management Following Major Gynecologic Surgery: Effect on Opioid Rescue, Return of Bowel Function, Cost and Length of Hospital Stay.
Brief Title: Efficacy of IV Acetaminophen for Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2013.08.22.F2
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Post-operative Pain
Keywords: IV Acetaminophen; Ofirmev; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Normal Saline) (Placebo Comparator): Morphine patient-controlled-anesthesia (PCA) for the initial 24 hours post-operation with a low-dose basal rate (0.5mg/hr) and patient administered boluses prn. Oral oxycodone from 24-48 hours post-operation will be used prn for pain and then patients will be transitioned to oral combined oxycodone/acetaminophen for the remainder of their hospital stay. Normal saline 100cc IV will be infused as placebo every 6 hours for a total of eight doses with the first dose being given at time of anesthesia induction.
  Interventions: Drug: Placebo
- Experimental (IV Acetaminophen) (Active Comparator): Morphine PCA for the initial 24 hours post-operation with low-dose basal rate (0.5mg/hr) with patient administered boluses prn. IV acetaminophen 1,000mg will be given every six hours for a total of eight doses with the first dose being given at time of anesthesia induction. Oral oxycodone from 24-48 hours post-operation will be used prn and then patients will be transitioned to oral combined oxycodone/acetaminophen for the remainder of their hospital stay.
  Interventions: Drug: IV acetaminophen

INTERVENTIONS:
Drug: Placebo — Normal saline (100cc) will be given IV as the placebo medication every six hours for a total of eight doses with the first dose being given at time of anesthesia induction.
  Other Names: IV Placebo
  Arms: Experimental (Normal Saline)
Drug: IV acetaminophen — IV acetaminophen (1,000mg) will be given every six hours for a total of eight doses with the first dose being given at time of anesthesia induction.
  Other Names: Ofirmev
  Arms: Experimental (IV Acetaminophen)

SUMMARY:
The investigators' goal in this planned prospective, randomized, patient blinded study is to compare our standard of care as the control group to an experimental group in which patients receive preemptive IV acetaminophen dosing that is continued every 6 hours for a total of 8 doses in patients who have undergone major gynecologic surgery. The outcomes analyzed will include amount of rescue opioids required, time to return of bowel function, length of hospital stay, and patient satisfaction. The hypothesis is that the addition of IV acetaminophen will decrease the need for opioid rescue and thereby decrease the incidence of associated gastrointestinal side effects including nausea, vomiting, bloating, and constipation. The hope is that it will affect the final outcome of quicker return of bowel function, increased patient satisfaction, shortened hospital stay and prove to be an overall more effective postoperative pain management approach.

DETAILED DESCRIPTION:
This is a patient-blinded prospective study in which patients that undergo major gynecologic surgery via an open abdominal approach will be randomized into two arms:

1. Control Group: Morphine patient-controlled-anesthesia (PCA) for the initial 24 hours post-operation with a low-dose basal rate (0.5mg/hr) and patient administered boluses prn. Oral oxycodone from 24-48 hours post-operation will be used prn for pain and then patients will be transitioned to oral combined oxycodone/acetaminophen for the remainder of their hospital stay. Normal saline 100cc IV will be infused as placebo every 6 hours for a total of eight doses with the first dose being given at time of anesthesia induction.
2. Experimental Group: Morphine PCA for the initial 24 hours post-operation with low-dose basal rate (0.5mg/hr) with patient administered boluses prn. IV acetaminophen 1,000mg will be given every six hours for a total of eight doses with the first dose being given at time of anesthesia induction. Oral oxycodone from 24-48 hours post-operation will be used prn and then patients will be transitioned to oral combined oxycodone/acetaminophen for the remainder of their hospital stay.

Outcomes that will be analyzed include the amount of opioids used; time to return of bowel function designated as passage of flatus; time to first bowel movement if it occurs while inpatient; duration of hospital stay; and patient symptoms and satisfaction at the 24 and 48 hour marks as well as at time of discharge.

ELIGIBILITY:
Inclusion Criteria:

-Female patients undergoing major gynecologic surgery via an open abdominal approach. The included surgeries would be exploratory laparotomy with or without removal of uterus, fallopian tubes, or ovaries.

Exclusion Criteria:

* Patients with baseline preoperative liver function enzymes (AST and ALT) that are greater than twice the upper limit of normal would be excluded.
* Patients with baseline CrCl <30.
* Patients that require intensive postoperative care and delayed extubation will typically require additional sedation which would impede adequate evaluation of the two study pain regimens as they are designed to be patient controlled.
* Patients with complications unrelated to the pain regimens that prolong their stay would be excluded from the evaluation of hospital stay and cost effectiveness analyses. Examples would include but are not limited to pre-renal azotemia and acute renal failure; pneumonia; venous thromboembolism; or need for re-exploration laparotomy.
* Allergy to acetaminophen would exclude those patients set to enter the experimental IV acetaminophen study arm. One exception would be if the allergy were trivial and related to route of administration such as mild nausea with oral acetaminophen.
* Patients that undergo a bowel resection during surgery as it may adversely effect return of bowel function
* Patients that have required regular opioid intake for the 7 days preceding surgery.
* NSAIDs within 8 hours of surgery.
* Chronic steroid use with the exception of low-dose inhaled steroid formulations.
* Chronic alcohol or drug abuse.
* Patients currently pregnant.
* Patients unable to provide informed consent.
* Age >85
* Any physical, medical, and mental condition that would make participation in the study inadvisable.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12-24 (Actual); Primary Completion 2014-06-04 (Actual); Study Completion 2014-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Randolph, DO, MS, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Health Foundation, Canton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 participants were enrolled between December 2013 and May 2014 at local institution
Groups:
- Experimental (Normal Saline): Placebo: Normal saline (100cc) will be given IV as the placebo medication every six hours for a total of eight doses with the first dose being given at time of anesthesia induction.
  Morphine patient-controlled-anesthesia (PCA) for the initial 24 hours post-operation with a low-dose basal rate (0.5mg/hr) and patient administered boluses prn. Oral oxycodone from 24-48 hours post-operation will be used prn for pain and then patients will be transitioned to oral combined oxycodone/acetaminophen for the remainder of their hospital stay.
- Experimental (IV Acetaminophen): IV acetaminophen: IV acetaminophen (1,000mg) will be given every six hours for a total of eight doses with the first dose being given at time of anesthesia induction.
  Morphine PCA for the initial 24 hours post-operation with low-dose basal rate (0.5mg/hr) with patient administered boluses prn. Oral oxycodone from 24-48 hours post-operation will be used prn and then patients will be transitioned to oral combined oxycodone/acetaminophen for the remainder of their hospital stay.
Period: Overall Study
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Started | 34 | 34
Completed | 29 | 30
Not Completed | 5 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Did not complete satisfaction surveys | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen) | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.34 (16.101) | 51.73 (12.690) | 51.05 (14.358)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Opioid Rescue - 48 Hours
Description: Mean number opioid rescue in the first 48 hours calculated by converting all opiates to intravenous morphine
Time Frame: First 48 hours including pre-operative and intra-operative medications
Measure: Mean (Standard Deviation); unit: Milligrams of intravenous morphine equiv
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 29 | 30
Milligrams of intravenous morphine equiv | 54.4803 (22.86841) | 48.9253 (22.94435)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority; p = .356, t-test for Equality of Means; Mean Difference (Final Values) = 5.55501, 95% CI 2-sided [-6.39040 to 17.50042], Standard Error of Mean 5.96535

2. Secondary Outcome: Return of Bowel Function
Description: Time to return of bowel function (passage of flatus) in hours
Time Frame: Duration of hospital stay (up to 7 days).
Population: Only participants with documented return of bowel function prior to discharge were analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 26 | 28
Hours | 68.0878 (22.99293) | 56.5696 (27.88443)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority; p = .105, t-test for Equality of Means; Median Difference (Final Values) = 11.51818, 95% CI 2-sided [-2.49963 to 25.53599], Standard Error of Mean 6.98569

3. Secondary Outcome: Patient Satisfaction - Pain Control at 24 Hours, 48 Hours, and Discharge
Description: Subjects will rate their overall satisfaction with pain control on a 5-point Likert scale: 1=Strongly disagree; 2=Disagree; 3=Neutral; 4=Agree; 5=Strongly Agree
Time Frame: At 24 hours 48 hours, and discharge (up to 7 days)
Population: Participants who completed the pain satisfaction survey at 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 24 | 26
score on a scale
  At 24 hours | 4.21 (.721) | 4.19 (1.021)
  At 48 hours | 4.08 (.881) | 4.04 (.824)
  At Discharge | 4.58 (.654) | 4.23 (.951)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority; p = .029, ANOVA

4. Secondary Outcome: Patient Satisfaction - Nausea Control at 24 Hours, 48 Hours, and Discharge
Description: Subjects will rate their overall satisfaction with nausea control on a 5-point Likert scale 1=Strongly disagree; 2=Disagree; 3=Neutral; 4=Agree; 5=Strongly Agree
Time Frame: At 24 hours, 48 Hours, and Discharge (up to 7 days)
Population: Participants who completed the nausea control survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 24 | 26
score on a scale
  At 24 hours | 3.88 (.900) | 3.73 (1.041)
  At 48 hours | 4.12 (.992) | 3.50 (1.068)
  At Discharge | 4.17 (.761) | 3.65 (.797)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority — Within subjects Analysis of Variance (ANOVA) of time, sphericity assumed, was used for pain, nausea, bloating and pruritus; p = .643, ANOVA

5. Secondary Outcome: Patient Satisfaction - Bloating at 24 Hours, 48 Hours, and Discharge
Description: Subjects will rate their overall satisfaction with bloating on a 5-point likert scale 1=Strongly disagree; 2=Disagree; 3=Neutral; 4=Agree; 5=Strongly Agree
Time Frame: At 24 hours, 48 Hours, and Discharge (up to 7 days)
Population: Participants who completed the bloating satisfaction survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 24 | 26
score on a scale
  At 24 hours | 3.58 (1.472) | 4.23 (.951)
  At 48 hours | 3.75 (1.152) | 3.69 (1.050)
  At Discharge | 3.79 (1.141) | 3.35 (1.093)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = .217, ANOVA

6. Secondary Outcome: Patient Satisfaction - Pruritis at 24 Hours, 48 Hours, and Discharge
Description: Subjects will rate their overall satisfaction with pruritis control on a 5-point likert scale 1=Strongly disagree; 2=Disagree; 3=Neutral; 4=Agree; 5=Strongly Agree
Time Frame: At 24 hours, 48 Hours, and Discharge (up to 7 days)
Population: Participants who completed the pruritus satisfaction survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 24 | 26
score on a scale
  At 24 hours | 3.71 (1.459) | 3.58 (1.391)
  At 48 hours | 3.67 (1.404) | 3.85 (1.120)
  At Discharge | 3.54 (1.382) | 3.88 (1.177)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = .647, ANOVA

7. Secondary Outcome: Length of Stay
Description: Mean length of post-operative stay in days
Time Frame: Surgery to discharge
Population: Participants experiencing adverse event leading to increased length of stay were not analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
Number analyzed (Participants) | 29 | 30
Days | 3.62 (1.147) | 3.57 (1.305)
Statistical Analysis 1: Comparison: Experimental (Normal Saline) vs Experimental (IV Acetaminophen); Test type: Superiority; Mean Difference (Final Values) = .054, 95% CI 2-sided [-.587 to .695], Standard Error of Mean .320

ADVERSE EVENTS:
Time Frame: Surgery to Discharge (up to 7 days)
Arm/Group | Experimental (Normal Saline) | Experimental (IV Acetaminophen)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 2/34 | 1/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (Normal Saline) (N=34) | Experimental (IV Acetaminophen) (N=34)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pain perception and tolerance is an individual characteristics that cannot be controlled. Other limitations include small sample size and reliance on participants to complete surveys at prescribed time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No